CLINICAL TRIAL: NCT05304715
Title: Bezlotoxumab Yielded Outcomes by Addressing Personalized Needs in Clostridioides Difficile Infection: The BEYOND Double-Blind Randomized Clinical Trial
Brief Title: Bezlotoxumab Yielded Outcomes by Addressing Personalized Needs in Clostridioides Difficile Infection
Acronym: BEYOND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BEYOND; 2021-005473-10 (EudraCT Number)
Record Dates: First submitted 2022-03-12; First posted 2022-03-31 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Clostridioides Difficile Infection; Stool Microbiome; Organ Dysfunction Syndrome; Clostridioides Difficile Infection Recurrence; Mortality
Keywords: Bezlotoxumab
MeSH Terms: conditions — Clostridium Infections | interventions — bezlotoxumab; Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a prospective, 1:1 randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patients will be treated with 250ml of normal saline 0.9% or 5% dextrose water as single intravenous infusion of one hour within 72 hours from the start of standard-of-care treatment. Standard-of-care treatment will be prescribed to all patients at the discretion of the attending physicians according to local guidelines or to their own decision.
  Interventions: Drug: Normal saline 0.9% or 5% dextrose water
- Bezlotoxumab (Active Comparator): Patients will be treated with bezlotoxumab at a dose of 10mg per kg of body weight (up to maximum of 1000mg) dissolved in 250ml of normal saline 0.9% or 5% dextrose water as single intravenous infusion of one hour within 72 hours from the start of standard-of-care treatment. Standard-of-care treatment will be prescribed to all patients at the discretion of the attending physicians according to local guidelines or to their own decision.
  Interventions: Drug: Bezlotoxumab

INTERVENTIONS:
Drug: Bezlotoxumab — Single intravenous infusion of bezlotoxumab
  Other Names: Standard-of-care treatment according to local guidelines or to the decision of the attending physicians.
  Arms: Bezlotoxumab
Drug: Normal saline 0.9% or 5% dextrose water — Single intravenous infusion - Placebo arm
  Other Names: Standard-of-care treatment according to local guidelines or to the decision of the attending physicians
  Arms: Placebo

SUMMARY:
Previous data have shown that integrated information from single nucleotide polymorphisms (SNPs) of the host DNA, interleukin 8 (IL-8) and the enrichment of the stool microbiome can indicate the patients with infection by Clostridioides difficile (CDI) who are at risk for unfavorable outcome. This integrated information is forming the BEYOND score. The aim of the BEYOND randomized clinical trial (RCT) is to investigate if adjunctive bezlotoxumab treatment to the current standard-of-care may decrease the likelihood of unfavorable outcome for patients who score positive by the BEYOND score.

DETAILED DESCRIPTION:
Clostridioides difficile infection (CDI) is an emerging infection with increased point-prevalence per year as reported both for the United States and for European countries. Current evidence suggests that CDI is a complex interaction between the host and the offending pathogen where physician intervention plays a pivotal role. Although originally conceived to be a hospital-acquired infection, it becomes more and more recognized that many cases are community-acquired. This underscores the significance of the host in the pathogenesis of CDI. CDI is traditionally considered to derive from the direct oral transmission from one host to the other in the hospital environment. However, a recent survey in three large hospitals in Wales analyzing the whole genome C.difficile isolated from 499 cases of diarrhea positive for glutamate dehydrogenase (GDH) revealed that the vast majority of isolates of C.difficile had different nucleotide sequences suggesting against the direct transmission from one patient to the other in the vast majority of cases. The complex interaction between the host and C.difficile ending to infection is modulated by environmental factors like antibiotic consumption, proton pump inhibitor intake and prolonged hospitalization.

The main endpoint of all randomized clinical trials (RCTs) of new antimicrobials targeting C.difficile is sustained clinical response that is defined as the composite of the resolution of the infection at the end of treatment without any CDI relapse within the first 40 days. This endpoint is mainly targeting to demonstrate if newly developed agents are superior over the comparator vancomycin in the minimization of relapse risk. However, recent data outscore the lack of substantial merit of this endpoint as many cases of CDI bear an intrinsic danger of unfavorable outcome without this being incorporated in the RCT endpoints. More precisely, a substantial rate of patients dies after the end of oral treatment between days 12 and 40 probably as a result of emerging organ dysfunction in the field of CDI colitis. Recent epidemiological data coming from the United States challenge even more the traditional way of our thinking of CDI. More precisely, in a prospective survey of 30,326 patients it was shown that the risk of unfavorable outcome and death was greater among first-time infected patients than in relapsed cases. This survey reports that mortality from the first CDI case may be as high as 28%. These cases of CDI associated with an unfavorable outcome leading to surgery and hospitalization in an intensive care unit are associated with a tremendous cost mounting to $34,149 per case. Surprisingly when data of the two registration RCTs of fidaxomicin were combined reduced CDI mortality was shown over the comparator vancomycin treatment. This observation strengthens the belief that the substantial merit of new agents is not in preventing CDI relapse but in saving lives.

The pivotal RCTs of fidaxomicin influenced the design of the MODIFY studies in a way that the inclusion criteria of these studies comprised not only cases of CDI infection of moderate severity but also patients with high chance of relapse. Half of the enrolled patient population was aged equal to or above 65 years and another quarter of enrolled patients had history of at least one episode of CDI. In these trials, patients with CDI receiving oral treatment with metronidazole, vancomycin or fidaxomicin were randomized to one single dose of adjunctive treatment with placebo or the monoclonal antibody targeting the toxin B of C.difficile bezlotoxumab, or the monoclonal antibody targeting the toxin A of C.difficile actoxumab or both antibodies. Results revealed that bezlotoxumab treatment reduced considerably the risk of relapse whereas the intake of actoxumab did not affect the clinical outcome of CDI. However, the efficacy of bezlotoxumab treatment on other variables of unfavorable outcome was not analyzed.

One main argument against new treatments targeting C.difficile is the substantial cost. This argument is based on the fact that there are no tools that can discriminate between patients at high risk for unfavorable outcome that are in need of new treatments from patients at low risk from unfavorable outcome that will benefit from standard-of-care vancomycin treatment.

In order to distinguish these patients, the investigators introduce a score which is called BEYOND. In this score, patients with CDI are at increased likelihood for unfavorable outcome if they meet any of the following:

1. Gene score for susceptibility to CDI more than 53. The score is provided by the following equation:

   (Carriage of C allele of rs12148744 x 27) - (carriage of C allele of rs714024 x 27) - (carriage of C allele of rs721059 x 29) + (carriage of T allele of rs4311028 x 33) - (carriage of A allele of rs62183547 x 25) + (carriage of C allele of rs1128266 x 12) - (carriage of T allele of rs4279595 x 17) + (carriage of G allele of rs175006 x 11) + (carriage of T allele of rs3859214 x 17) + (carriage of G allele of rs7222870 x 15) - (carriage of G allele of rs5086600 x 9) + (carriage of T allele of rs7240534 x 12) + (carriage of G allele of rs20911172 x 11) - (carriage of C allele of rs17680671 x 17) OR
2. Score provided by the following equation more than 9:

   [Hemoglobin <9.5 g/dl x 10] + [serum urea >64.5 mg/dl x 14] + [serum interleukin-8 >227 pg/ml x 19] - [carriage of G allele of rs2091172 x 17] OR
3. More than 3log10 of gammaproteobacteria or Enterobacteriaceae or Enterobacteriales in the stool

ELIGIBILITY:
Inclusion Criteria:

1. Age equal to or above18 years.
2. Both genders.
3. Written informed consent provided by the patient or by their legal representative in case of patients unable to consent.
4. In case of non-menopausal women, unwillingness to become pregnant during the study period. Women of child-bearing potential will be screened by a urine pregnancy test before inclusion in the study.
5. Diarrhea defined as at least 3 episodes of unformed stool in the past 24hours.
6. Positive stool for C.difficile. This is defined as any stool sample positive for the presence of glutamate dehydrogenase (GDH) and for the presence of toxin A and/or B.
7. Positive BEYOND score i.e. meeting any of the following:

Gene score for susceptibility to CDI more than 53. The score is provided by the following equation:

(Carriage of C allele of rs12148744 x 27) - (carriage of C allele of rs714024 x 27) - (carriage of C allele of rs721059 x 29) + (carriage of T allele of rs4311028 x 33) - (carriage of A allele of rs62183547 x 25) + (carriage of C allele of rs1128266 x 12) - (carriage of T allele of rs4279595 x 17) + (carriage of G allele of rs175006 x 11) + (carriage of T allele of rs3859214 x 17) + (carriage of G allele of rs7222870 x 15) - (carriage of G allele of rs5086600 x 9) + (carriage of T allele of rs7240534 x 12) + (carriage of G allele of rs20911172 x 11) - (carriage of C allele of rs17680671 x 17) OR

Score provided by the following equation more than 9:

[Hemoglobin <9.5 g/dl x 10] + [serum urea >64.5 mg/dl x 14] + [serum interleukin-8 >227 pg/ml x 19] - [carriage of G allele of rs2091172 x 17] OR More than 3log10 of gammaproteobacteria or Enterobacteriaceae or Enterobacteriales in the stool

Exclusion Criteria:

* Age below 18 years
* Denial for written informed consent
* Known allergy to bezlotoxumab
* Pregnancy or lactation. Women of child-bearing potential will be screened by a urine pregnancy test before inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2023-06-04 (Actual); Study Completion 2023-06-04 (Actual)

PRIMARY OUTCOMES:
Comparison of bezlotoxumab over placebo on reducing the incidence of progression into organ dysfunction defined as any increase of the baseline total SOFA score by at least 2 points. | 40 days
  Progression into organ dysfunction is defined as any increase of the baseline total SOFA score by at least 2 points. Need for colectomy or admission in the Intensive Care Unit counts also as organ dysfunction.
Comparison of bezlotoxumab over placebo on reducing the incidence of relapse of Clostridioides difficile infection | 40 days
  Relapse is defined as the return of more than three unformed bowel movements in 24 hours with a positive stool toxin test necessitating retreatment
Comparison of bezlotoxumab over placebo on reducing the incidence of death | 40 days
  Death

SECONDARY OUTCOMES:
Comparison of bezlotoxumab over placebo regarding the time to first organ dysfunction | 1-40 days
  This is defined as the presentation of organ dysfunction in any of the enrolled patients of each group starting from the day of blind allocation until Day 40.
Comparison of bezlotoxumab over placebo regarding the time to relapse of CDI | 1-40 days
  The relapse of CDI is under daily follow-up until Day 40. Relapse is defined as the return of more than three unformed bowel movements in 24 hours with a positive stool toxin test necessitating retreatment.
Comparison of bezlotoxumab over placebo regarding survival time | 1-40 days
  Survival until Day 40 from study enrolment
Comparison of bezlotoxumab over placebo regarding overall cost of hospitalization | 1-40 days
  This is calculated starting from the day of blind allocation until Day 40
Validation of the BEYOND score | 1-40 days
  This is done by comparing the incidence of the primary endpoint between patients who have failed screening in the trial and patients who were enrolled in the trial and who were allocated to the placebo arm. Positive BEYOND score is expected to be associated with worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos J Giamarellos-Bourboulis, MD, PhD, Study Chair — Hellenic Sepsis Study Group
Locations (11):
- Greece (11):
  - 2nd Department of Internal Medicine, University General Hospital of Alexandroupolis, Alexandroupoli
  - 1st Department of Internal Medicine, THRIASIO General Hospital of Eleusis, Athens
  - 2nd Department of Internal Medicine, Thriasio General Hospital, Athens
  - 1st University Department of Internal Medicine, LAIKO General Hospital of Athens,, Athens
  - 1st University Department of Propaedeutic Surgery, IPPOKRATEION General Hospital, Athens
  - 4th Department of Internal Medicine, Attikon University Hospital, Athens
  - 1st Department of Internal Medicine, General University Hospital of Ioannina, Ioannina
  - Department of Internal Medicine, Larissa University Hospital, Larissa
  - Department of Internal Medicine, University General Hospital of Patras PANAGIA I VOITHIA, Pátrai
  - 2nd Department of Internal Medicine, Tzanneion General Hospital, Piraeus
  - 1st Department of Internal Medicine, AHEPA University General Hospital of Thessaloniki, Thessaloniki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Psarrakis C, Tziolos NR, Matzarakis V, Kumar V, Stylianakis E, Sidiropoulou C, Tasouli E, Iliopoulou K, Samarkos M, Metallidis S, Georgiadou S, Akinosoglou K, Bolanou A, Hatziagelaki E, Kostaki A, Panagopoulos P, Toutouzas K, Milionis H, Adamis G, Poulakou G, Lada M, Skoutelis A, Alexiou Z, Symbardi S, Chrysos G, Netea MG, Giamarellos-Bourboulis EJ. A randomized controlled trial of precision bezlotoxumab treatment for Clostridioides difficile infection. Cell Rep Med. 2026 Jan 20;7(1):102533. doi: 10.1016/j.xcrm.2025.102533. Epub 2026 Jan 2. PMID 41483804